CLINICAL TRIAL: NCT01877824
Title: Consequences of Fast-track Training in Surgery in Denmark in Selected Operative Skills.
Brief Title: Study of Fast-track Surgery in Hernia Repair and Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); Aalborg University Hospital (Other); TRYG Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MEDU001
Record Dates: First submitted 2013-05-27; First posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Surgical Training
Keywords: Surgery; Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast-track training (Experimental): A skills-lap course (1 day) followed by opportunity to perform 20 planned surgical procedures of each type (open groin hernia repair and laparoscopic cholecystectomy) under supervision and within 4-8 weeks. Videorecording at start, mid and end and at follow-up before ending first year of training.
  Interventions: Other: Fast-track training
- Control (No Intervention): Follows the existing training program without intervention. Video recording of the trainee performing a open groin hernia repair and a laparoscopic cholecystectomy procedure at start end end of first training year.

INTERVENTIONS:
Other: Fast-track training
  Arms: Fast-track training

SUMMARY:
All Danish trainees in surgery in a two-year period asked for participation when enrolled in the formal five-year training program for specialty in surgery. The participants are randomized for either educational intervention or control (without intervention). The intervention group receive a skills-lab course in hernia repair followed by an opportunity to perform 20 groin hernia repairs in their departments within 4-8 weeks. Their performance will be video recorded three times during the intervention and as follow-up at end of the first year of training. After termination of the hernia training program a similar program for laparoscopic cholecystectomies are made. Each participant receive both intervention. The control group are video recorded at start of their first year and at end. All videos are blindly assessed with a validated rating scale of operative performance. The purpose is to assess if a fast-track program improves technical skills and if a change is sustained. Furthermore we want to compare outcome in similar training programs in open and laparoscopic skills.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors accepted for formal surgical training in Denmark in 2010-11.

Exclusion Criteria:

* Current experience in surgery exceeding need of supervision in groin hernia and cholecystectomy procedures.
* Employed at a non-participating hospital.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Technical skills in performed surgical procedures | Three years
  Blinded video recordings of the trainees' performances are rated with a validated rating scale of technical skills.

SECONDARY OUTCOMES:
Operative time | Three years
  The time in performing the surgical procedures are recorded.
Satisfaction | Three years
  The intervention group participants are asked for their experience and satisfaction with a fast-track program

CONTACTS AND LOCATIONS:
Overall Officials: Peder Charles, MD, DMSci, Study Chair — University of Aarhus
Locations (1):
- Centre of Medical Education, Aarhus, Denmark

REFERENCES:
- [Derived] Carlsen CG, Lindorff-Larsen K, Funch-Jensen P, Lund L, Konge L, Charles P. Module based training improves and sustains surgical skills: a randomised controlled trial. Hernia. 2015 Oct;19(5):755-63. doi: 10.1007/s10029-015-1357-6. Epub 2015 Mar 3. PMID 25731946